CLINICAL TRIAL: NCT01960517
Title: A Feasibility Assessment of a New Urinary Catheter: The Alternative Catheter System ACS)
Brief Title: Feasibility Assessment of ACS Catheter
Acronym: ACS1
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor decision not to proceed with study
Sponsor: Alternative Urological Catheter Systems Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AUCS/2013/ACS01
Record Dates: First submitted 2013-10-07; First posted 2013-10-10 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2013-10

CONDITIONS: Urological
Keywords: Urinary; Incontinence; Catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Catheter placed (Experimental)
  Interventions: Device: ACS Catheter

INTERVENTIONS:
Device: ACS Catheter

SUMMARY:
This is a single centre, non-randomised, baseline controlled, prospective pilot clinical trial to be undertaken at Rotherham General Hospital, Rotherham, UK.

The study will examine the safety and performance of a new urinary catheter, the Alternative Catheter System (ACS) (Alternative Urological Catheter Systems Ltd (AUCS), Bristol, UK) which has been developed to reduce the morbidity of long-term catheterisation and the acknowledged deficiencies of the conventional Foley urinary catheter.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age.
2. Patient or authorised representative must be able to comprehend and sign the Informed Consent Form prior to enrolment in the study.
3. Capable of using a catheter valve to empty the bladder and able to communicate their experience with the system OR who has a carer able to fulfil these tasks.
4. Fitted with a suprapubic catheter (at least 2 weeks post insertion).
5. Ability to attend out-patient clinic at regular intervals throughout the study and able to participate for a maximum of 8 weeks.
6. History of catheter blockages, bypassing or episodes of pyrexia and bacteraemia in the last 2 months.

Exclusion Criteria:

1. <18 years of age.
2. Pregnant or lactating females.
3. History of catheter associated septicaemia in the past month.
4. Evidence of current systemic infection.
5. Bladder pathology such as a tumour or stone >0.5cm as determined by cystoscopy.
6. Flaccid bladder.
7. BMI>35.
8. Current participation in another device or drug study.
9. Unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Retention of the ACS catheter | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mr Isa Idhem, Principal Investigator — Rotherham NHS Foundation Trust
Locations (1):
- Rotherham NHS Foundation Trust, Rotherham General Hospital, Rotherham, United Kingdom